CLINICAL TRIAL: NCT00761579
Title: An Open-Label Prospective, Non-Comparative Study To Explore The Tolerability, Safety and Effectiveness Upon Transition to Paliperidone Slow-Release Tablet in Schizophrenic Patients
Brief Title: Paliperidone Extended Release(ER) Effectiveness Study to Evaluate the Objective Symptom Change and Symptomatic Remission
Acronym: PERFECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015250; PAL-KOR-4002
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Antipsychotics Agents
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone (Experimental): Paliperidone oral tablet was administered once daily at a starting dose of either 3 milligram (mg), 6 mg or 9 mg for 48 weeks, wherein recommended dose was 6 mg and dose range was 3 to 12 mg per day.
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone oral tablet was administered once daily at a starting dose of either 3 milligram (mg), 6 mg or 9 mg for 48 weeks, wherein recommended dose was 6 mg and dose range was 3 to 12 mg per day.
  Other Names: R076477; Invega Slow-Release Tablet

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of flexibly dosed paliperidone extended-release (ER) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label, prospective (study following participants forward in time), single arm, and non-comparative study of paliperidone Extended Release(ER) in participants with schizophrenia (after switching from the existing drug to paliperidone ER). The total study duration will be approximately of 48 weeks per participant. The study consists of 2 parts: Screening (that is, 14 days before study commences on Day 1); Treatment (single-oral dose of paliperidone for 48 weeks, dose ranging from 3 to 12 milligram). Efficacy of the participants will primarily be evaluated by Positive and Negative Syndrome Scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Childbearing potential women who consent to the use of the consistently permissible contraception (oral contraceptive, contraceptive injection, intrauterine device, double barrier method and contraceptive patch)
* Participants who are compliant with self-medication or can receive consistent help or support
* Participants who need to change the antipsychotic drug to another one for the following reasons among the participants treated with an antipsychotic drug for more than two weeks before the screening (1) Group of lack of efficacy: the antipsychotic drug is clinically required to be changed because there is no or little therapeutic response despite the appropriately dosed antipsychotic therapy (2) Group of lack of tolerance: the antipsychotic drug is required to be changed due to lack of tolerance to the existing antipsychotic drug or the safety issue (3) Group of lack of compliance: the antipsychotic drug is required to be changed due to lack of medication compliance or the participant wants to change the antipsychotic drug)
* Have schizophrenia diagnosis by Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)

Exclusion Criteria:

* Participants with the past history of neuroleptic malignant syndrome (NMS)
* Participants who are suspicious of having clinically significant risk including suicide or aggressive behavior and are expected to unable to complete the study(based on the investigator's judgment)
* Participants with severe preexisting gastrointestinal narrowing (pathologic or iatrogenic) or participants who cannot swallow the drug whole (the study drug must not be chewed, divided, melted or grinded because it can impact the study drug release profile)
* Participants with significant abnormal findings in blood chemistry, hematological and urine analyses which are clinically significant at the investigator's discretion
* Female Participants who are pregnant or are breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (8):
- South Korea (8):
  - Busan
  - Chunjoo
  - Daegu
  - Goyang-si
  - Ilsan
  - Kyounggi
  - Kyunggi-Do
  - Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone: Paliperidone oral tablet was administered once daily at a starting dose of either 3 milligram (mg) for 48 weeks, wherein recommended dose was 6 mg and dose range was 3 to 12 mg per day.
Period: Overall Study
Arm/Group | Paliperidone
Started | 190
Completed | 98
Not Completed | 92
Not completed — Adverse Event | 10
Not completed — Death | 2
Not completed — Lack of Efficacy | 21
Not completed — Lost to Follow-up | 16
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 34
Not completed — Lack of compliance | 2
Not completed — Protocol deviation | 1
Not completed — Drug overdose | 1
Not completed — Aggravation of depression | 1
Not completed — Aggravation of symptoms by changing drug | 1
Not completed — Lost survey form | 1
Not completed — Intake of prohibited concomitant drug | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 97
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
  Units on a scale | 79.42 (19.64)
Positive and Negative Syndrome Scale (PANSS) - Positive Subscale Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS Positive Subscale assesses seven positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
  Units on a scale | 18.96 (6.19)
Positive and Negative Syndrome Scale (PANSS) - Negative Subscale Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS Negative Subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
  Units on a scale | 20.61 (5.97)
Positive and Negative Syndrome Scale (PANSS) - General Psychopathology Subscale Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS General Psychopathology Subscale Score assesses 16 general psychopathology symptoms. The symptoms are rated on a 7-point scale, with a range of 16 (absent) to 112 (extreme psychopathology).
  Units on a scale | 18.00 (5.56)
Personal and Social Performance Scale (PSP) Score [Mean (Standard Deviation); unit: Units on a scale] — The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty).
  Units on a scale | 54.08 (14.84)
Drug Attitude Inventory (DAI-10) [Mean (Standard Deviation); unit: Units on a scale] — DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10.
  Units on a scale | 3.01 (4.31)
Subjective Well-being Under Neuroleptic (SWN-20) Scale Score [Mean (Standard Deviation); unit: Units on a scale] — The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood.
  Units on a scale | 73.64 (16.87)
Daytime Drowsiness [Mean (Standard Deviation); unit: Units on a scale] — Daytime Drowsiness was assessed by an 11-point visual analog scale. Participants indicated on the 11-point visual analog scale (score ranging from 0 to 100 millimeter) how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time). Scores were averaged for the previous 7 days.
  Units on a scale | 45.65 (29.97)
Sleep Quality [Mean (Standard Deviation); unit: Units on a scale] — Sleep quality was assessed by an 11-point visual analog scale. Participants indicated on the 11-point visual analog scale (score ranging from 0 to 100 millimeter) how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time). Scores were averaged for the previous 7 days.
  Units on a scale | 61.90 (27.73)
Symptom Checklist 90-R (SCL90-R) [Mean (Standard Deviation); unit: Units on a scale] — The SCL90-R (Derogatis, 1992) measures 9 domains, including somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, which provides a global index of distress, the Global Severity Index (GSI). SCL-90-R includes 90 items rated on 5-point scale, ranging from 0 (not at all) to 4 (extremely). Total scale score range from 0 to 360. Higher scores indicate worsening of disease.
  Units on a scale | 91.72 (65.10)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 48
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening. Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: Intent to treat (ITT) population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone ER: Lack of Efficacy: Paliperidone ER tablet in dose range of 3 to 12 milligram (mg) per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy (switching of antipsychotic drug was clinically necessary because of no or insufficient response to treatment despite antipsychotic drug therapy at an adequate dose).
- Paliperidone ER: Lack of Tolerability: Paliperidone ER tablet in dose range of 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of tolerability (switching of antipsychotic drug was necessary due to lack of tolerability in the existing antipsychotic drug).
- Paliperidone ER: Lack of Compliance: Paliperidone ER tablet in dose range of 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of compliance (switching of antipsychotic drug was necessary due to lack of compliance in the existing antipsychotic drug).
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 144 | 21 | 25
Units on a scale | 11.57 (16.95) | 6.43 (13.94) | 16.36 (17.44)

2. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Positive Subscale Score at Week 48
Description: The PANSS Positive Subscale assesses seven positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology). Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 144 | 21 | 25
Units on a scale | 3.53 (5.23) | 1.05 (2.75) | 5.00 (6.40)

3. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Negative Subscale Score at Week 48
Description: The PANSS Negative Subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology). Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 144 | 21 | 25
Units on a scale | 2.53 (4.60) | 2.19 (4.07) | 3.36 (5.51)

4. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - General Psychopathology Subscale Score at Week 48
Description: The PANSS General Psychopathology Subscale Score assesses 16 general psychopathology symptoms. The symptoms are rated on a 7-point scale, with a range of 16 (absent) to 112 (extreme psychopathology). Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 144 | 21 | 25
Units on a scale | 5.51 (9.41) | 3.19 (8.68) | 8.00 (8.30)

5. Secondary Outcome: Change From Baseline in Personal and Social Performance Scale (PSP) Score at Week 48
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty). Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 144 | 21 | 25
Units on a scale | -6.73 (14.16) | -2.38 (9.86) | -11.36 (13.90)

6. Secondary Outcome: Change From Baseline in Drug Attitude Inventory (DAI-10) at Week 48
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10, higher score indicates positive SR (compliant) and lower score indicates negative SR (non-compliant). Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 140 | 21 | 24
Units on a scale | -0.01 (4.72) | -0.95 (4.27) | 0.08 (4.19)

7. Secondary Outcome: Change From Baseline in Subjective Well-being Under Neuroleptic (SWN-20) Scale Score at Week 48
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 140 | 21 | 25
Units on a scale | -1.17 (14.37) | -5.05 (14.03) | 2.40 (11.85)

8. Secondary Outcome: Change From Baseline in Daytime Drowsiness at Week 48
Description: Daytime Drowsiness was assessed by an 11-point visual analog scale. Participants indicated on the 11-point visual analog scale (score ranging from 0 to 100 millimeter) how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time). Scores were averaged for the previous 7 days. Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 140 | 21 | 25
millimeter (mm) | 5.40 (34.11) | 2.10 (27.76) | 11.40 (24.61)

9. Secondary Outcome: Change From Baseline in Sleep Quality at Week 48
Description: Sleep quality was assessed by an 11-point visual analog scale. Participants indicated on the 11-point visual analog scale (score ranging from 0 to 100 millimeter) how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time). Scores were averaged for the previous 7 days. Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 140 | 21 | 25
millimeter (mm) | 1.50 (32.94) | -7.76 (31.20) | 3.40 (35.34)

10. Secondary Outcome: Change From Baseline in Symptom Checklist 90-R (SCL90-R) at Week 48
Description: The SCL90-R (Derogatis, 1992) measures 9 domains, including somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, which provides a global index of distress, the Global Severity Index (GSI). SCL-90-R includes 90 items rated on 5-point scale, ranging from 0 (not at all) to 4 (extremely). Total scale score range from 0 to 360. Higher scores indicate worsening of disease. Total scale score range from 0 to 360. Higher scores indicate worsening of disease. Change from Baseline is calculated as value at Baseline minus value at Week 48. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability | Paliperidone ER: Lack of Compliance
Number analyzed (Participants) | 140 | 21 | 25
Units on a scale | 14.88 (48.32) | 12.38 (32.01) | 25.44 (44.41)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Description: Safety population included all the eligible participants who received paliperidone extended-release (ER) at least once .
Arm/Group | Paliperidone
Serious Adverse Events (participants affected / at risk) | 23/190
Other Adverse Events (participants affected / at risk) | 109/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=190)
Inguinal Hernia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Agitated Depression (Psychiatric disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Completed Suicide (Psychiatric disorders) | 2
Confusional State (Psychiatric disorders) | 1
Depressive Symptom (Psychiatric disorders) | 2
Hallucination, Auditory (Psychiatric disorders) | 1
Persecutory Delusion (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 6
Suicidal Behaviour (Psychiatric disorders) | 1
Suicide Attempt (Psychiatric disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=190)
Hyperprolactinaemia (Endocrine disorders) | 11
Vision Blurred (Eye disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Dry Mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 7
Gait Disturbance (General disorders) | 5
Weight Decreased (Investigations) | 5
Weight Increased (Investigations) | 29
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 14
Akathisia (Nervous system disorders) | 35
Bradykinesia (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 8
Dysarthria (Nervous system disorders) | 5
Dyskinesia (Nervous system disorders) | 5
Dystonia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 4
Sedation (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 13
Amenorrhoea (Reproductive system and breast disorders) | 7

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less